CLINICAL TRIAL: NCT04575584
Title: A Phase 2/3, Randomized, Placebo-Controlled, Double-Blind Clinical Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of MK-4482 in Hospitalized Adults With COVID-19
Brief Title: Efficacy and Safety of Molnupiravir (MK-4482) in Hospitalized Adult Participants With COVID-19 (MK-4482-001)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4482-001; MK-4482-001 (Other: Merck); PHRR201210-003189 (Registry Identifier: PHRR); jRCT2031200404 (Registry Identifier: jRCT); 2020-003367-26 (EudraCT Number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — molnupiravir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Molnupiravir 200 mg (Experimental): 200 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Molnupiravir
- Part 1: Molnupiravir 400 mg (Experimental): 400 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Molnupiravir
- Part 1: Molnupiravir 800 mg (Experimental): 800 mg molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Molnupiravir
- Part 1: Placebo (Placebo Comparator): Placebo matching molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Placebo
- Part 2: Molnupiravir (Experimental): Molnupiravir (dose to be selected) administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Molnupiravir
- Part 2: Placebo (Placebo Comparator): Placebo matching molnupiravir administered orally every 12 hours for 5 days (10 doses total)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Molnupiravir — Molnupiravir administered orally in capsule form every 12 hours for 5 days (10 doses total)
  Arms: Part 1: Molnupiravir 200 mg; Part 1: Molnupiravir 400 mg; Part 1: Molnupiravir 800 mg; Part 2: Molnupiravir
Drug: Placebo — Placebo matching molnupiravir administered orally in capsule form every 12 hours for 5 days (10 doses total)
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
This study aims to evaluate the safety, tolerability and efficacy of molnupiravir (MK-4482) compared to placebo. The primary hypothesis is that molnupiravir is superior to placebo as assessed by the rate of sustained recovery through Day 29.

DETAILED DESCRIPTION:
This study was intended to include two parts: Part 1 was a dose-ranging phase 2 study, and Part 2 was a phase 3 study to evaluate the dose selected in Part 1. However, this study was terminated due to business reasons prior to conducting Part 2. Participants in Part 1 were followed until Month 7.

ELIGIBILITY:
Inclusion Criteria:

* Has documentation of polymerase chain reaction (PCR)-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection with sample collection ≤ 10 days prior to the day of randomization. PCR is the preferred method; however other diagnostic methods are allowed if authorized by use in the country
* Had initial onset of signs/symptoms attributable to COVID-19 for ≤10 days prior to the day of randomization and ≥1 sign/symptom attributable to COVID-19 present at randomization
* Requires medical care in the hospital for ongoing clinical manifestations of COVID-19 (not just for public health or quarantine purposes)
* Has mild, moderate, or severe COVID-19
* Is willing and able to take oral medication
* Males agree to the following during the intervention period and for at least 90 days after the last dose of study intervention: Refrain from donating sperm; and either abstain from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or must agree to use contraception
* Females are not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of child bearing potential (WOCBP); or is a WOCBP and using a contraceptive method that is highly effective (a low user dependency method OR a user dependent method in combination with barrier method), or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) for 28 days from the start of study intervention; a WOCBP must have a negative highly sensitive pregnancy test (serum test is required) within 24 hours before the first dose of study intervention

Exclusion Criteria:

* Has critical COVID-19 with any of the following: respiratory failure (including endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula (flow rates >20L/min with fraction of delivered oxygen ≥ 0.5), noninvasive positive pressure ventilation, or extracorporeal membrane oxygenation (ECMO))
* Is on dialysis or has reduced estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m^2 by the Modification of Diet in Renal Disease (MDRD) equation
* Has any of the following conditions: human immunodeficiency virus (HIV) with a recent viral load >50 copies/mL or cluster of differentiation 4 (CD4) <200 cell/mm^3; chemotherapy required within 6 weeks before randomization; a neutrophilic granulocyte absolute count <500/mm^3; autologous or allogeneic hematopoietic stem cell transplant recipient
* Has history of Hepatitis B or Hepatitis C infection with any of the following: 1) cirrhosis 2) end-stage liver disease 3) hepatocellular carcinoma 4) aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times the upper limit of normal at screening
* Has a history of acute pancreatitis within 3 months prior to randomization or a history of chronic pancreatitis
* Is taking or is anticipated to require any prohibited therapies
* Is unwilling to abstain from participating in another interventional clinical trial through Day 29 with an investigational compound or device, including those for COVID-19 therapeutics
* Is anticipated to require transfer to a non-study hospital within 72 hours
* Has a baseline heart rate of < 50 beats per minute at rest
* Has a platelet count <100,000/μL or received a platelet transfusion in the 5 days prior to randomization
* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments including but not limited to: participants who are not expected to survive longer than 48 hours after randomization or participants who are expected to require mechanical ventilation within 48 hours after randomization or participants with a recent history of mechanical ventilation or participants with conditions that could limit gastrointestinal absorption of capsule contents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (89):
- United States (20):
  - Kaiser Foundation Hospital - South Bay ( Site 1832), Harbor City, California
  - Cedars-Sinai Medical Center ( Site 1822), Los Angeles, California
  - University of California Davis Health ( Site 1809), Sacramento, California
  - University Of Florida ( Site 1810), Gainesville, Florida
  - Wellstar Kennestone Hospital ( Site 1801), Marietta, Georgia
  - Loretto Hospital ( Site 1838), Chicago, Illinois
  - LSU-HSC Shreveport ( Site 1824), Shreveport, Louisiana
  - Henry Ford Health System ( Site 1821), Detroit, Michigan
  - University of Mississippi Medical Center ( Site 1846), Jackson, Mississippi
  - University of Nebraska Medical Center ( Site 1835), Omaha, Nebraska
  - University of New Mexico, Health Sciences Center ( Site 1806), Albuquerque, New Mexico
  - Carolinas Medical Center ( Site 1850), Charlotte, North Carolina
  - ECU Adult Specialty Care ( Site 1865), Greenville, North Carolina
  - Sanford Health ( Site 1851), Fargo, North Dakota
  - Temple University ( Site 1836), Philadelphia, Pennsylvania
  - CHRISTUS Institute for Innovation & Advanced Clinical Care ( Site 1864), Corpus Christi, Texas
  - Houston Methodist Hospital ( Site 1863), Houston, Texas
  - Swedish Medical Center ( Site 1812), Edmonds, Washington
  - Valley Medical Center ( Site 1815), Renton, Washington
  - Swedish Medical Center ( Site 1861), Seattle, Washington
- Brazil (5):
  - Chronos Pesquisa Clínica ( Site 0105), Brasília, Federal District
  - Santa Casa de Misericordia de Belo Horizonte ( Site 0100), Belo Horizonte, Minas Gerais
  - Hospital de Clinicas da Universidade Federal do Parana ( Site 0104), Curitiba, Paraná
  - Hospital Tacchini ( Site 0107), Bento Gonçalves, Rio Grande do Sul
  - FUNFARME Hospital de Base Centro Integrado de Pesquisa ( Site 0101), São José do Rio Preto, São Paulo
- University Health Network - Toronto General Hospital ( Site 0201), Toronto, Ontario, Canada
- Chile (5):
  - Clinica Universidad de los Andes ( Site 0301), Santiago, Region M. de Santiago
  - Hospital Sotero del Rio [Santiago, Chile] ( Site 0304), Santiago, Region M. de Santiago
  - Complejo Hospitalario San Jose ( Site 0306), Santiago, Region M. de Santiago
  - Servicio de Salud Sur Hospital Lucio Cordova ( Site 0305), Santiago, Region M. de Santiago
  - Hospital Clinico Fusat ( Site 0300), Rancagua, Región del Libertador General Bernardo O’Higgins
- Colombia (6):
  - Hospital Pablo Tobon Uribe ( Site 0404), Medellín, Antioquia
  - Clinica de la Costa Ltda. ( Site 0402), Barranquilla, Atlántico
  - Hospital Universitario San Ignacio ( Site 0401), Bogotá, Bogota D.C.
  - Oncomedica S.A. ( Site 0406), Montería, Departamento de Córdoba
  - Fundacion Cardiovascular de Colombia ( Site 0403), Bucaramanca, Santander Department
  - Fundacion Valle del Lili ( Site 0400), Cali, Valle del Cauca Department
- France (6):
  - Groupe Hospitalier Pellegrin ( Site 0511), Bordeaux, Gironde
  - C.H.U. de Toulouse. Hopital de Purpan ( Site 0501), Toulouse, Midi-Pyrenees
  - Centre Hospitalier de Tourcoing ( Site 0502), Tourcoing, Nord
  - CHU Hopital Saint Antoine ( Site 0505), Paris
  - Hopital Bichat - Claude Bernard ( Site 0503), Paris
  - Pitie Salpetriere University Hospital-Infectious Disease - Tropical Diseases ( Site 0504), Paris, Île-de-France Region
- Israel (3):
  - Rambam Medical Center ( Site 2102), Haifa
  - Hadassah Medical Center. Ein Kerem ( Site 2103), Jerusalem
  - Chaim Sheba Medical Center ( Site 2100), Ramat Gan
- ASST Fatebenefratelli-Ospedale Sacco ( Site 0601), Milan, Italy
- Mexico (4):
  - Hospital Regional de Alta Especialidad del Bajio ( Site 0807), León, Guanajuato
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0800), Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0802), Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez ( Site 0803), Monterrey, Nuevo León
- Philippines (2):
  - University of the Philippines-Philippine General Hospital ( Site 0900), Manila, National Capital Region
  - Lung Center of the Philippines ( Site 0902), Quezon City, National Capital Region
- Poland (4):
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie ( Site 1004), Lublin, Lublin Voivodeship
  - Centrum Medyczne Pratia, Mazowiecki Szpital Specjalistyczny, Oddział Obserwacyjno - Zakaźny ( Site 1, Ostrołęka, Masovian Voivodeship
  - Centrum Medyczne w Lancucie Sp.zo.o. ( Site 1000), Łańcut, Podkarpackie Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. dr. Wladyslawa Bieganskiego ( Site 1001), Lodz-Baluty, Łódź Voivodeship
- Russia (8):
  - City Clinical Hospital #40 ( Site 1109), Moscow, Moscow
  - FSBI Central Hospital with Policlinics ( Site 1105), Moscow, Moscow
  - Moscow Clinical Hospital #52 ( Site 1103), Moscow, Moscow
  - Krasnogorsk City Hospital Number 1 ( Site 1119), Krasnogorsk, Moscow Oblast
  - City Hospital #40 ( Site 1113), Saint Petersburg, Sankt-Peterburg
  - City Pokrovskaya hospital ( Site 1116), Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital #1 ( Site 1112), Smolensk, Smolensk Oblast
  - Republican Clinical Infectious Hospital n.a. A.F. Agafonov ( Site 1100), Kazan', Tatarstan, Respublika
- South Africa (4):
  - IATROS International ( Site 1202), Bloemfontein, Free State
  - Wits Baragwanath Clinical Trial Site ( Site 1204), Soweto, Gauteng
  - TREAD Research ( Site 1201), Cape Town, Western Cape
  - Clinical Projects Research Centre ( Site 1205), Worcester, Western Cape
- South Korea (3):
  - Chungnam National University Hospital ( Site 2202), Daejeon, Taejon-Kwangyokshi
  - Inha University Hospital ( Site 2204), Incheon
  - The Catholic University of Korea Eunpyeong St Mary s Hospital ( Site 2205), Seoul
- Spain (6):
  - Hospital Universitari Vall d Hebron ( Site 1305), Barcelona, Catalonia
  - Hospital Clinic ( Site 1304), Barcelona
  - Hospital Universitari Germans Trias i Pujol ( Site 1303), Barcelona
  - Hospital Universitario Gregorio Maranon ( Site 1302), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 1301), Madrid
  - Hospital Universitario La Paz ( Site 1300), Madrid
- Ukraine (8):
  - Ivano-Frankivsk Regional Clinical Infectious Diseases Hospital ( Site 1605), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - CNE Central city clinical hospital of Ivano-Frankivsk city council ( Site 1604), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - MNE Ivano-Frankivsk Regional Phthisiology-Pulmonology Center ( Site 1603), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - CNPE of Kharkiv RC Regional Clinical Infectious Diseases Hospital ( Site 1606), Kharkiv, Kharkivs’ka Oblast’
  - Сommunal non-com. Institution Oleksandrivska clinical hospital Kyiv ( Site 1600), Kyiv, Kyivska Oblast
  - Odesa City Clinical Infectious Hospital ( Site 1611), Odesa, Odesa Oblast
  - Communal Non-Commercial Enterprise Central City Hospital ( Site 1615), Rivne, Rivne Oblast
  - Volyn Regional Clinical Hospital ( Site 1613), Lutsk, Volyn Oblast
- United Kingdom (3):
  - Royal Free London NHS Foundation Trust ( Site 1700), London, London, City of
  - King's College Hospital ( Site 1705), London, London, City of
  - North Manchester General Hospital ( Site 1701), Manchester

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Arribas JR, Bhagani S, Lobo SM, Khaertynova I, Mateu L, Fishchuk R, Park WY, Hussein K, Kim SW, Ghosn J, Brown ML, Zhang Y, Gao W, Assaid C, Grobler JA, Strizki J, Vesnesky M, Paschke A, Butterton JR, De Anda C. Randomized Trial of Molnupiravir or Placebo in Patients Hospitalized with Covid-19. NEJM Evid. 2022 Feb;1(2):EVIDoa2100044. doi: 10.1056/EVIDoa2100044. Epub 2021 Dec 16. PMID 38319178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 86 study centers in 15 countries.
Period: Overall Study
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Started | 75 | 75 | 76 | 78 | 0 (Study terminated prior to initiating Part 2) | 0 (Study terminated prior to initiating Part 2)
Treated | 73 | 73 | 72 | 75 | 0 | 0
Completed | 61 | 60 | 63 | 70 | 0 | 0
Not Completed | 14 | 15 | 13 | 8 | 0 | 0
Not completed — Death | 6 | 4 | 6 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 9 | 5 | 3 | 0 | 0
Not completed — Not recorded | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in Part 2 arms due to early study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo | Total
Number analyzed (Participants) | 75 | 75 | 76 | 78 | 0 | 0 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (14.2) | 57.0 (14.0) | 56.8 (13.7) | 57.1 (14.2) |  |  | 57.0 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 32 | 34 | 0 | 0 | 132
  Male | 43 | 41 | 44 | 44 | 0 | 0 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 32 | 28 | 27 | 0 | 0 | 114
  Not Hispanic or Latino | 47 | 42 | 46 | 49 | 0 | 0 | 184
  Unknown or Not Reported | 1 | 1 | 2 | 2 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 1 | 2 | 0 | 0 | 6
  Asian | 10 | 8 | 4 | 1 | 0 | 0 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 4 | 6 | 7 | 0 | 0 | 18
  White | 58 | 52 | 54 | 63 | 0 | 0 | 227
  More than one race | 6 | 7 | 9 | 5 | 0 | 0 | 27
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time-to-sustained Recovery
Description: The median time to sustained recovery is reported. Sustained recovery is defined as 1) the participant is alive and not hospitalized; or 2) the participant is alive and medically ready for discharge as determined by the investigator.
Time Frame: Up to 29 days
Population: All randomized participants in Part 1 who received ≥1 dose of study drug are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
days | 9.0 [7.0 to 10.0] | 9.0 [8.0 to 10.0] | 9.0 [8.0 to 11.0] | 9.0 [8.0 to 11.0] |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5620, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.68 to 1.45] — Based on Cox regression model with Efron's method of tie handling
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.3145, Log Rank; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.78 to 1.65] — Based on Cox regression model with Efron's method of tie handling
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.4894, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.69 to 1.47] — Based on Cox regression model with Efron's method of tie handling

2. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: The number of participants with at least 1 AE is presented. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 19 days (during treatment and 14-day follow-up)
Population: All randomized participants in Part 1 who received ≥1 dose of study drug are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants | 40 | 36 | 45 | 46 |  |

3. Primary Outcome: Number of Participants Who Discontinued Study Intervention Due to an AE
Description: The number of participants discontinuing from study treatment due to an AE is presented. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 5 days
Population: All randomized participants in Part 1 who received ≥1 dose of study drug are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants | 0 | 1 | 0 | 0 |  |

4. Secondary Outcome: Number of Participants With All-cause Mortality
Description: The number of participants with all-cause mortality through Day 29 is presented. All-cause mortality is defined as death due to any cause. Any participants with an unknown survival status at Day 29 were imputed as deceased.
Time Frame: Up to 29 days
Population: All randomized participants in Part 1 who received ≥1 dose of study drug are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants | 4 | 5 | 4 | 1 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.1642, Miettinen and Nurminen method; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [-2.3 to 12.1] — Miettinen and Nurminen method. Unknown Day 29 survival status treated as failure
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.0900, Miettinen and Nurminen method; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [-1.1 to 13.9] — Miettinen and Nurminen method. Unknown Day 29 survival status treated as failure
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.1594, Miettinen and Nurminen method; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [-2.3 to 12.3] — Miettinen and Nurminen method. Unknown Day 29 survival status treated as failure

5. Secondary Outcome: Odds of a More Favorable Response on Pulmonary Ordinal Outcome Score on Day 3
Description: Pulmonary score is a score on an ordinal scale which focuses on respiratory sequalae based on oxygen requirements using 7 mutually exclusive categories. The score ranges from 1 ("can independently undertake personal usual activities with minimal or no symptoms") to 7 ("death") with a higher score indicating more severe respiratory sequalae. The number of participants at each score category is presented.
Time Frame: Day 3
Population: All randomized participants in Part 1 who received ≥1 dose of study drug and have data available at the relevant time point are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  1 | 25 | 20 | 21 | 16 |  |
  2: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  2 | 2 | 7 | 0 | 7 |  |
  3: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  3 | 21 | 20 | 23 | 25 |  |
  4: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  4 | 16 | 16 | 19 | 14 |  |
  5: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  5 | 7 | 9 | 6 | 10 |  |
  6: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  6 | 1 | 0 | 3 | 1 |  |
  7: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  7 | 0 | 0 | 0 | 0 |  |
  Missing | 1 | 1 | 0 | 2 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.3623, Wald Chi-Square; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.73 to 2.35] — Based on the proportional odds model with Pulmonary score categories as the response variable. Due to sparse data, the final model includes only treatment as covariate. Confidence intervals (CIs) are based on Wald Chi-Square Test
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5714, Wald Chi-Square; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.66 to 2.12] — Based on the proportional odds model with Pulmonary score categories as the response variable. Due to sparse data, the final model includes only treatment as covariate. CIs are based on Wald Chi-Square Test
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.9313, Wald Chi-Square; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.54 to 1.75] — [estimate comment as in outcome 5, analysis 2]

6. Secondary Outcome: Odds of a More Favorable Response on Pulmonary Ordinal Outcome Score on End of Treatment (EOT [Day 5])
Description: as for outcome 5
Time Frame: EOT (Day 5)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  1 | 30 | 22 | 26 | 27 |  |
  2: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  2 | 6 | 5 | 4 | 4 |  |
  3: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  3 | 17 | 18 | 15 | 16 |  |
  4: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  4 | 10 | 14 | 14 | 14 |  |
  5: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  5 | 7 | 8 | 8 | 8 |  |
  6: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  6 | 1 | 1 | 3 | 1 |  |
  7: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  7 | 0 | 0 | 0 | 0 |  |
  Missing | 2 | 5 | 2 | 5 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.4398, Wald Chi-Square; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.70 to 2.30] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.6277, Wald Chi-Square; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.47 to 1.57] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.7069, Wald Chi-Square; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.49 to 1.62] — [estimate comment as in outcome 5, analysis 2]

7. Secondary Outcome: Odds of a More Favorable Response on Pulmonary Ordinal Outcome Score on Day 10
Description: as for outcome 5
Time Frame: Day 10
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  1 | 44 | 39 | 33 | 38 |  |
  2: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  2 | 4 | 4 | 4 | 5 |  |
  3: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  3 | 8 | 8 | 14 | 10 |  |
  4: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  4 | 5 | 7 | 8 | 10 |  |
  5: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  5 | 4 | 3 | 5 | 4 |  |
  6: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  6 | 3 | 0 | 3 | 3 |  |
  7: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  7 | 0 | 3 | 0 | 0 |  |
  Missing | 5 | 9 | 5 | 5 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.2422, Wald Chi-Square; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.77 to 2.85] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.4789, Wald Chi-Square; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.66 to 2.44] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.6052, Wald Chi-Square; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.45 to 1.59] — [estimate comment as in outcome 5, analysis 2]

8. Secondary Outcome: Odds of a More Favorable Response on Pulmonary Ordinal Outcome Score on Day 15
Description: as for outcome 5
Time Frame: Day 15
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  1 | 45 | 44 | 41 | 42 |  |
  2: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  2 | 7 | 2 | 2 | 5 |  |
  3: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  3 | 6 | 6 | 14 | 10 |  |
  4: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  4 | 3 | 5 | 3 | 6 |  |
  5: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  5 | 2 | 1 | 0 | 4 |  |
  6: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  6 | 4 | 1 | 7 | 3 |  |
  7: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  7 | 0 | 3 | 1 | 1 |  |
  Missing | 6 | 11 | 4 | 4 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.2644, Wald Chi-Square; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.75 to 2.88] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.2184, Wald Chi-Square; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.77 to 3.14] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.9771, Wald Chi-Square; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.53 to 1.94] — [estimate comment as in outcome 5, analysis 2]

9. Secondary Outcome: Odds of a More Favorable Response on Pulmonary Ordinal Outcome Score on Day 29
Description: as for outcome 5
Time Frame: Day 29
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  1 | 46 | 47 | 47 | 49 |  |
  2: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  2 | 2 | 2 | 2 | 5 |  |
  3: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  3 | 4 | 5 | 9 | 7 |  |
  4: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  4 | 5 | 1 | 3 | 5 |  |
  5: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  5 | 0 | 0 | 0 | 0 |  |
  6: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  6 | 2 | 0 | 5 | 2 |  |
  7: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  7 | 4 | 4 | 3 | 1 |  |
  Missing | 10 | 14 | 3 | 6 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.9945, Wald Chi-Square; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.46 to 2.06] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.3227, Wald Chi-Square; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.67 to 3.37] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5200, Wald Chi-Square; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.39 to 1.61] — [estimate comment as in outcome 5, analysis 2]

10. Secondary Outcome: Odds of a More Favorable Response on Pulmonary+ Ordinal Outcome Score on Day 3
Description: Pulmonary+ score is a score on an ordinal scale which is a 7-category assessment that captures the range of disease severity in hospitalized participants, including coagulation-related complications and respiratory dysfunction. The score ranges from 1 ("can independently undertake personal usual activities with minimal or no symptoms") to 7 ("death") with a higher score indicating more severe respiratory sequalae. The number of participants at each score category is presented.
Time Frame: Day 3
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  1 | 25 | 20 | 21 | 16 |  |
  2: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  2 | 2 | 7 | 0 | 7 |  |
  3: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  3 | 20 | 20 | 23 | 25 |  |
  4: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  4 | 16 | 16 | 19 | 14 |  |
  5: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  5 | 7 | 9 | 6 | 10 |  |
  6: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  6 | 2 | 0 | 3 | 1 |  |
  7: number analyzed (Participants) | 72 | 72 | 72 | 73 | 0 | 0
  7 | 0 | 0 | 0 | 0 |  |
  Missing | 1 | 1 | 0 | 2 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.4472, Wald Chi-Square; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.70 to 2.25] — Based on the proportional odds model with Pulmonary+ score categories as the response variable. Due to sparse data, the final model includes only treatment as covariate. CIs are based on Wald Chi-Square Test
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5714, Wald Chi-Square; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.66 to 2.12] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.9313, Wald Chi-Square; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.54 to 1.75] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Odds of a More Favorable Response on Pulmonary+ Ordinal Outcome Score on EOT (Day 5)
Description: as for outcome 10
Time Frame: EOT (Day 5)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  1 | 30 | 22 | 26 | 27 |  |
  2: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  2 | 6 | 5 | 4 | 4 |  |
  3: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  3 | 16 | 18 | 15 | 16 |  |
  4: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  4 | 10 | 14 | 14 | 14 |  |
  5: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  5 | 7 | 8 | 8 | 8 |  |
  6: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  6 | 2 | 1 | 3 | 1 |  |
  7: number analyzed (Participants) | 71 | 68 | 70 | 70 | 0 | 0
  7 | 0 | 0 | 0 | 0 |  |
  Missing | 2 | 5 | 2 | 5 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5222, Wald Chi-Square; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.67 to 2.21] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.6277, Wald Chi-Square; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.47 to 1.57] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.7069, Wald Chi-Square; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.49 to 1.62] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Odds of a More Favorable Response on Pulmonary+ Ordinal Outcome Score on Day 10
Description: as for outcome 10
Time Frame: Day 10
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  1 | 44 | 39 | 33 | 38 |  |
  2: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  2 | 4 | 4 | 4 | 5 |  |
  3: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  3 | 8 | 8 | 14 | 10 |  |
  4: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  4 | 4 | 7 | 8 | 10 |  |
  5: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  5 | 4 | 3 | 4 | 4 |  |
  6: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  6 | 4 | 0 | 4 | 3 |  |
  7: number analyzed (Participants) | 68 | 64 | 67 | 70 | 0 | 0
  7 | 0 | 3 | 0 | 0 |  |
  Missing | 5 | 9 | 5 | 5 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.2627, Wald Chi-Square; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.75 to 2.80] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.4789, Wald Chi-Square; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.66 to 2.44] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5938, Wald Chi-Square; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.45 to 1.58] — [estimate comment as in outcome 10, analysis 1]

13. Secondary Outcome: Odds of a More Favorable Response on Pulmonary+ Ordinal Outcome Score on Day 15
Description: as for outcome 10
Time Frame: Day 15
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  1 | 45 | 44 | 41 | 42 |  |
  2: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  2 | 7 | 2 | 2 | 5 |  |
  3: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  3 | 6 | 6 | 14 | 10 |  |
  4: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  4 | 3 | 5 | 3 | 6 |  |
  5: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  5 | 2 | 1 | 0 | 4 |  |
  6: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  6 | 4 | 1 | 7 | 3 |  |
  7: number analyzed (Participants) | 67 | 62 | 68 | 71 | 0 | 0
  7 | 0 | 3 | 1 | 1 |  |
  Missing | 6 | 11 | 4 | 4 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.2644, Wald Chi-Square; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.75 to 2.88] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.2184, Wald Chi-Square; Odds Ratio (OR) = 1.55, 95% CI 2-sided [0.77 to 3.14] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.9771, Wald Chi-Square; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.53 to 1.94] — [estimate comment as in outcome 10, analysis 1]

14. Secondary Outcome: Odds of a More Favorable Response on Pulmonary+ Ordinal Outcome Score on Day 29
Description: as for outcome 10
Time Frame: Day 29
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  1: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  1 | 46 | 47 | 47 | 49 |  |
  2: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  2 | 2 | 2 | 2 | 5 |  |
  3: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  3 | 4 | 5 | 9 | 7 |  |
  4: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  4 | 5 | 1 | 3 | 5 |  |
  5: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  5 | 0 | 0 | 0 | 0 |  |
  6: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  6 | 2 | 0 | 5 | 2 |  |
  7: number analyzed (Participants) | 63 | 59 | 69 | 69 | 0 | 0
  7 | 4 | 4 | 3 | 1 |  |
  Missing | 10 | 14 | 3 | 6 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.9445, Wald Chi-Square; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.46 to 2.06] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.3227, Wald Chi-Square; Odds Ratio (OR) = 1.50, 95% CI 2-sided [0.67 to 3.37] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5200, Wald Chi-Square; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.39 to 1.61] — [estimate comment as in outcome 10, analysis 1]

15. Secondary Outcome: Odds of a More Favorable Response in the Clinical Risk of Mortality Category From the National Early Warning Score
Description: The National Early Warning Score (Royal College of Physicians, 2012) assesses a participant's degree of illness as assessed by clinical risk prediction categories based on a set of vital sign measurements. There are 7 physiological parameters: respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, and temperature. A score of 0 to 3 was allocated to each parameter except supplemental oxygen use (score of 0 [no] or 2 [yes]) and level of consciousness (score of 0 or 3 with 0 = normal health condition and 3 = worst health condition). All scores were summed to get an aggregate score. Aggregate NEWS score ranged from 0 to 19, with higher scores meaning more severity/higher risk: low risk (score 0 to 4); low to medium risk (score of 3 in any individual parameter); medium risk (score 5 to 6); high risk (score 7 to 19). The number of participants at each aggregate risk category is presented.
Time Frame: EOT (Day 5)
Population: All randomized participants in Part 1 who received ≥1 dose of study drug and have data at the relevant time point are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  Low: number analyzed (Participants) | 70 | 64 | 69 | 69 | 0 | 0
  Low | 57 | 45 | 52 | 55 |  |
  Medium: number analyzed (Participants) | 70 | 64 | 69 | 69 | 0 | 0
  Medium | 8 | 8 | 9 | 11 |  |
  High: number analyzed (Participants) | 70 | 64 | 69 | 69 | 0 | 0
  High | 5 | 11 | 8 | 3 |  |
  Missing: number analyzed (Participants) | 70 | 64 | 69 | 69 | 0 | 0
  Missing | 3 | 9 | 3 | 6 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.8732, Wald Chi-Square; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.46 to 2.47] — Proportional odds model with National Early Warning Score (NEWS) categories as the response variable. Due to sparse data, the final model includes only treatment as covariate. CIs are based on Wald Chi-Square Test
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.1277, Wald Chi-square; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.25 to 1.19] — Proportional odds model with NEWS categories as the response variable. Due to sparse data, the final model includes only treatment as covariate. CIs are based on Wald Chi-Square Test
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.4326, Wald Chi-Square; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.33 to 1.61] — [estimate comment as in outcome 15, analysis 2]

16. Secondary Outcome: Odds of a More Favorable Response on WHO 11-point Ordinal Outcomes Score on a Scale on Day 3
Description: The World Health Organization (WHO) outcome scale is an 11-point ordinal score that categorizes clinical progression. Score ranges from 0 ("uninfected") to 10 ("dead") with higher score indicating clinical progression. The number of participants at each score category is presented.
Time Frame: Day 3
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  0 | 0 | 0 | 0 | 0 |  |
  1 | 0 | 0 | 0 | 0 |  |
  2 | 1 | 1 | 0 | 2 |  |
  3 | 1 | 0 | 0 | 1 |  |
  4 | 27 | 27 | 21 | 24 |  |
  5 | 36 | 36 | 42 | 37 |  |
  6 | 7 | 9 | 6 | 10 |  |
  7 | 0 | 0 | 0 | 0 |  |
  8 | 0 | 0 | 2 | 0 |  |
  9 | 1 | 0 | 1 | 1 |  |
  10 | 0 | 0 | 0 | 0 |  |
  Missing | 0 | 0 | 0 | 0 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.6830, Wald Chi-Square; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.50 to 2.88] — Based on the proportional odds model with WHO-11 score categories as the response variable. Due to sparse data, the final model includes only treatment as covariate. CIs are based on Wald Chi-Square Test
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 1.000, Wald Chi-Square; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.42 to 2.39] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.8244, Wald Chi-Square; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.37 to 2.20] — [estimate comment as in outcome 16, analysis 1]

17. Secondary Outcome: Odds of a More Favorable Response on WHO 11-point Ordinal Outcomes Score on a Scale on EOT (Day 5)
Description: as for outcome 16
Time Frame: EOT (Day 5)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  0: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  0 | 2 | 0 | 1 | 0 |  |
  1: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  1 | 2 | 1 | 1 | 2 |  |
  2: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  2 | 3 | 5 | 0 | 9 |  |
  3: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  3 | 0 | 2 | 2 | 1 |  |
  4: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  4 | 29 | 20 | 27 | 25 |  |
  5: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  5 | 27 | 31 | 28 | 26 |  |
  6: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  6 | 7 | 8 | 8 | 8 |  |
  7: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  7 | 0 | 0 | 0 | 0 |  |
  8: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  8 | 1 | 1 | 1 | 0 |  |
  9: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  9 | 0 | 0 | 2 | 1 |  |
  10: number analyzed (Participants) | 71 | 68 | 70 | 72 | 0 | 0
  10 | 0 | 0 | 0 | 0 |  |
  Missing | 2 | 5 | 2 | 3 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5022, Wald Chi-Square; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.36 to 1.64] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.5204, Wald Chi-Square; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.37 to 1.64] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.0991, Wald Chi-Square; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.24 to 1.13] — [estimate comment as in outcome 16, analysis 1]

18. Secondary Outcome: Odds of a More Favorable Response on WHO 11-point Ordinal Outcomes Score on a Scale on Day 10
Description: as for outcome 16
Time Frame: Day 10
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  0: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  0 | 3 | 4 | 2 | 3 |  |
  1: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  1 | 10 | 7 | 7 | 7 |  |
  2: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  2 | 26 | 19 | 22 | 21 |  |
  3: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  3 | 3 | 4 | 7 | 8 |  |
  4: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  4 | 8 | 16 | 7 | 13 |  |
  5: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  5 | 11 | 9 | 14 | 11 |  |
  6: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  6 | 4 | 2 | 5 | 3 |  |
  7: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  7 | 0 | 0 | 1 | 0 |  |
  8: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  8 | 2 | 0 | 0 | 3 |  |
  9: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  9 | 1 | 0 | 2 | 0 |  |
  10: number analyzed (Participants) | 68 | 64 | 67 | 69 | 0 | 0
  10 | 0 | 3 | 0 | 0 |  |
  Missing | 5 | 9 | 5 | 6 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.6346, Wald Chi-Square; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.60 to 2.29] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.7596, Wald Chi-Square; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.46 to 1.75] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.8879, Wald Chi-Square; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.49 to 1.84] — [estimate comment as in outcome 16, analysis 1]

19. Secondary Outcome: Odds of a More Favorable Response on WHO 11-point Ordinal Outcomes Score on a Scale on Day 15
Description: as for outcome 16
Time Frame: Day 15
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  0: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  0 | 10 | 8 | 10 | 8 |  |
  1: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  1 | 12 | 12 | 9 | 11 |  |
  2: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  2 | 25 | 25 | 27 | 27 |  |
  3: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  3 | 7 | 5 | 4 | 8 |  |
  4: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  4 | 4 | 3 | 3 | 5 |  |
  5: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  5 | 4 | 4 | 7 | 4 |  |
  6: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  6 | 2 | 0 | 0 | 3 |  |
  7: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  7 | 0 | 0 | 2 | 1 |  |
  8: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  8 | 3 | 0 | 1 | 0 |  |
  9: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  9 | 0 | 1 | 4 | 2 |  |
  10: number analyzed (Participants) | 67 | 61 | 68 | 70 | 0 | 0
  10 | 0 | 3 | 1 | 1 |  |
  Missing | 6 | 12 | 4 | 5 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.6002, Wald Chi-Square; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.55 to 2.82] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.4733, Wald Chi-Square; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.58 to 3.21] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.6220, Wald Chi-Square; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.38 to 1.78] — [estimate comment as in outcome 16, analysis 1]

20. Secondary Outcome: Odds of a More Favorable Response on WHO 11-point Ordinal Outcomes Score on a Scale on Day 29
Description: as for outcome 16
Time Frame: Day 29
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
Number analyzed (Participants) | 73 | 73 | 72 | 75 | 0 | 0
Participants
  0: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  0 | 25 | 17 | 29 | 22 |  |
  1: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  1 | 4 | 13 | 7 | 9 |  |
  2: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  2 | 24 | 21 | 17 | 24 |  |
  3: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  3 | 3 | 2 | 7 | 7 |  |
  4: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  4 | 0 | 2 | 0 | 0 |  |
  5: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  5 | 1 | 0 | 0 | 4 |  |
  6: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  6 | 0 | 0 | 0 | 0 |  |
  7: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  7 | 0 | 0 | 2 | 0 |  |
  8: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  8 | 2 | 0 | 2 | 2 |  |
  9: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  9 | 0 | 0 | 1 | 0 |  |
  10: number analyzed (Participants) | 63 | 59 | 68 | 69 | 0 | 0
  10 | 4 | 4 | 3 | 1 |  |
  Missing | 10 | 14 | 4 | 6 |  |
Statistical Analysis 1: Comparison: Part 1: Molnupiravir 200 mg vs Part 1: Placebo; Test type: Superiority; p = 0.7871, Wald Chi-Square; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.28 to 2.60] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 2: Comparison: Part 1: Molnupiravir 400 mg vs Part 1: Placebo; Test type: Superiority; p = 0.9598, Wald Chi-Square; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.31 to 3.06] — [estimate comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: Part 1: Molnupiravir 800 mg vs Part 1: Placebo; Test type: Superiority; p = 0.6670, Wald Chi-Square; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.27 to 2.31] — [estimate comment as in outcome 16, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: All randomized participants are included in the all-cause mortality assessment; only confirmed (no imputed) deaths are reported.
  All participants who received ≥1 dose of study treatment are included in the assessment of serious adverse events (SAEs) and nonserious AEs.
Arm/Group | Part 1: Molnupiravir 200 mg | Part 1: Molnupiravir 400 mg | Part 1: Molnupiravir 800 mg | Part 1: Placebo | Part 2: Molnupiravir | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 6/75 | 4/75 | 7/76 | 2/78 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 11/73 | 9/73 | 13/72 | 12/75 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 11/73 | 11/73 | 7/72 | 13/75 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Molnupiravir 200 mg (N=73) | Part 1: Molnupiravir 400 mg (N=73) | Part 1: Molnupiravir 800 mg (N=72) | Part 1: Placebo (N=75) | Part 2: Molnupiravir (N=0) | Part 2: Placebo (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Physical deconditioning (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | NA | NA
COVID-19 (Infections and infestations) | 7 (7) | 4 (4) | 5 (5) | 6 (6) | NA | NA
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | NA | NA
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | NA | NA
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | NA | NA
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | NA | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | NA | NA
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Molnupiravir 200 mg (N=73) | Part 1: Molnupiravir 400 mg (N=73) | Part 1: Molnupiravir 800 mg (N=72) | Part 1: Placebo (N=75) | Part 2: Molnupiravir (N=0) | Part 2: Placebo (N=0)
Constipation (Gastrointestinal disorders) | 5 (5) | 2 (2) | 0 (0) | 5 (5) | NA | NA
Alanine aminotransferase increased (Investigations) | 4 (4) | 5 (5) | 7 (7) | 8 (8) | NA | NA
Aspartate aminotransferase increased (Investigations) | 3 (3) | 5 (5) | 5 (6) | 3 (3) | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 0 (0) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT04575584/Prot_SAP_000.pdf